CLINICAL TRIAL: NCT02486900
Title: Real-time fMRI Neurofeedback as a Treatment Tool for Alcohol Dependence
Brief Title: Neurofeedback & Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, David Linden, Professor of Translational Neuroscience, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRAINTRAINAD
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Alcohol Dependence
Keywords: Craving; Cue Reactivity; Neurofeedback
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurofeedback training group (Experimental): The neurofeedback group will perform 6 training sessions over a period of 4 months: 4 fortnightly sessions in the first two months will be followed by 2 monthly 'booster' sessions. Each session will include several behavioural assessments and fMRI-based neurofeedback training in an MRI scanner (1 h). The neurofeedback training phase will be be followed-up by two behavioural assessments 8 and 12 months after the first training.
  Interventions: Device: fMRI-based neurofeedback
- Treatment-as-usual control group (No Intervention): The control group will receive treatment as usual (e.g. medication, counselling) but no neurofeedback training during the study period. Patients in the control group will be invited for four behavioural assessment sessions (baseline assessment, follow-up assessments 4/8/12 months after baseline).

INTERVENTIONS:
Device: fMRI-based neurofeedback — During scanning patients will be exposed to picture stimuli (showing alcoholic drinks and life goals) projected on a screen behind the scanner and viewed through a mirror attached on the MRI head coil. In each session patients will be trained to down-regulate/up-regulate activation levels in brain areas that show reliable responses to the alcohol/life goals pictures in a 'localiser' scan. Self-regulation of these brain responses will then be guided by real-time feedback of alcohol/life goals-cue elicited activation, consisting of changes in the visible alcohol/life goals picture (decreasing size = successful down-regulation; increasing size = successful upregulation). Functional MRI data will be acquired in short blocks having a duration of 5-8 minutes.
  Arms: Neurofeedback training group

SUMMARY:
The study aims to examine whether the neurofeedback method (based on functional magnetic resonance imaging [fMRI]) can help patients with alcohol dependence to control their urges to drink alcohol and thus to remain abstinent. Potential effects of neurofeedback on abstinence and drinking behaviour will be evaluated based on the comparison between a group of patients receiving multiple sessions of neurofeedback training and a group of patients receiving treatment as usual over the same period of time.

DETAILED DESCRIPTION:
Neurofeedback is a non-invasive neuroscientific tool in which participants receive real-time feedback about their brain activity while undergoing functional magnetic resonance imaging. Previous research has shown that participants can successfully use the feedback to self-regulate their brain responses. In this study patients who have successfully completed a detoxification programme will be trained to down-regulate/upregulate responses of motivational brain regions that are activated during exposure to alcohol/life goal-related stimuli (pictures of alcoholic drinks/life goals related). The investigators hypothesise that learning to self-regulate these neural responses will enable patients to better control craving responses to environmental alcohol cues after detoxification treatment. Patients in the intervention group will undergo 6 neurofeedback training sessions, spread across 4 months. Outcomes of the training will be compared with a group of patients who will not do the neurofeedback training but receive standard treatment (e.g. support groups and medication).

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of detoxification programme within a time window of 1 to 6 months before the recruitment
* Abstinence since detoxification treatment

Exclusion Criteria:

* Ongoing regular abuse of illicit substances except cannabis
* History of psychotic disorders not related to alcohol
* IQ < 70
* Involvement in other interventional research in the past 6 months
* MRI counter-indications, e.g. claustrophobia, pregnancy, active medical implants, passive implants deemed unsuitable, metallic dust in the eyes, certain types of metal prostheses, surgical clips, previous experience with metalworking without eye protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Indices of drinking (continuous) - % days abstinent | 4 months after baseline assessment/first training
  Derived from the Timeline Followback Calendar.
Indices of drinking (continuous) - drinks per drinking day | 4 months after baseline assessment/first training
  Derived from the Timeline Followback Calendar.
Indices of drinking (continuous) - % days of 'heavy drinking' | 4 months after baseline assessment/first training
  Defined as 8 or more alcohol units per day/men or 6 or more units/women. Derived from the Timeline Followback Calendar.

SECONDARY OUTCOMES:
Drinking urges/craving assessed with the Drinking Urges Questionnaire (DUQ) | Assessed 4 months, 8 months and 12 months after baseline
Drinking urges/craving assessed with the Obsessive Compulsive Drinking Scale (OCDS) | Assessed 4 months, 8 months and 12 months after baseline
Drinking urges/craving (attentional bias) assessed with the alcohol stroop test | Assessed 4 months, 8 months and 12 months after baseline
Craving self-ratings during scanning (neurofeedback group only) | Assessed 2, 4, 6, 8, 12, 16 weeks after baseline (each training session)
Profile of Mood States Questionnaire | Assessed 4 months, 8 months and 12 months after baseline
Beck Depression Inventory | Assessed 4 months, 8 months and 12 months after baseline
Hospital Anxiety and Depression Scale | Assessed 4 months, 8 months and 12 months after baseline
NHS Resource Use Questionnaire | Assessed 4 months, 8 months and 12 months after baseline
Debriefing Questionnaire (neurofeedback group only) | Assessed 2, 4, 6, 8, 12, 16 weeks after baseline (each training session)

CONTACTS AND LOCATIONS:
Overall Officials: David Linden, MD, Principal Investigator — Cardiff University
Locations (1):
- School of Medicine, Cardiff University, Cardiff, Wales, United Kingdom

REFERENCES:
- [Derived] Cox WM, Subramanian L, Linden DE, Luhrs M, McNamara R, Playle R, Hood K, Watson G, Whittaker JR, Sakhuja R, Ihssen N. Neurofeedback training for alcohol dependence versus treatment as usual: study protocol for a randomized controlled trial. Trials. 2016 Oct 3;17(1):480. doi: 10.1186/s13063-016-1607-7. PMID 27716290